CLINICAL TRIAL: NCT03872622
Title: Intestinal Response Patterns to Microbial Signals in the Healthy Rural & Urban and in the Crohn's Disease Host Gut
Brief Title: Intestinal Response Patterns to Microbial Signals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other); Washington University School of Medicine (Other); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Prof. Shomron BenHorin, Prof. Shomron Ben Horin, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5484-18-SMC
Record Dates: First submitted 2018-11-14; First posted 2019-03-13 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: CD - Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD patients (Other): New onset Crohn's disease patients
  Interventions: Other: Blood tests, intestinal biopsies, stool samples, environmental exposure questionnaire and FFQ questionnaire
- Healthy controls (Other): Patients' family members and healthy subjects undergoing colonoscopy for non-research purposes
  Interventions: Other: Blood tests, intestinal biopsies, stool samples, environmental exposure questionnaire and FFQ questionnaire

INTERVENTIONS:
Other: Blood tests, intestinal biopsies, stool samples, environmental exposure questionnaire and FFQ questionnaire — Blood tests, intestinal biopsies, stool samples, environmental exposure questionnaire and FFQ questionnaire.

SUMMARY:
A cohort of CD patients (total n=300) and a cohort of controls (healthy individuals and family members of CD patients, total n=200) will be recruited.

We will analyze gut host pattern of tissue immune system and epithelial responses to putative exposome and microbial triggers, expression data in the gut using mRNA expression studies and genetic analysis of the resident bacterial flora are necessary to identify specific molecules and signal pathways as well as specific bacterial taxa involved in aberrant response and instigation of inflammation that is the driver of Crohn's disease. Therefore, We will obtain stool & blood samples and intestinal biopsy and/or resection specimens from CD patients, and blood, stool and intestinal biopsy samples from healthy individuals and a-symptomatic family relatives undergoing colonoscopy for reasons un-related to the study (e.g screening colonoscopy).

Patients from both cohorts will also undergo environmental and dietary exposure survey. For environmental exposure, we will use the questionnaire developed by the International Organization of IBD (IOIBD), with some modification. Questions relate to five main different areas: (i) Childhood factors up to 20 years; (ii) food habits including daily, weekly or less frequent consumption; (iii) smoking habits; (iv) sanitary conditions such as the availability of in-house water tap, hot water tap or flush toilet; and (v) others factors including physical activity, oral contraceptive pill and stressful events before diagnosis.

For mapping dietary habits we will employ an interview conducted by a trained dietician and using the validated structured FFQ (Food frequency Questionnaire).

DETAILED DESCRIPTION:
Only adults>18YO will be included, Two cohorts will be included: A cohort of CD patients (including specific sub-cohorts of recruited known & new-onset CD and travelling CD patients and archived pathological specimens of post-operative CD, total n=300) and a cohort of controls (healthy individuals and family members of CD patients, total n=200). We will obtain stool & blood samples and intestinal biopsy and/or resection specimens from CD patients, and blood, stool and intestinal biopsy samples from healthy individuals and a-symptomatic family relatives undergoing colonoscopy for reasons un-related to the study (e.g screening colonoscopy).

After signing informed consent, Stool sample and blood sample (20cc) will be obtained. Enteric infections will be excluded by stool cultures, parasites including entameba, and C. difficile assay. Inflammatory markers (CRP in blood, calprotectin in stool) will be tested. Blood samples will undergo immune characterization including in vitro testing by immune cell activation, cytokine secretion measurements and cell-surface markers analysis by FACS. Two fecal samples per donor, (≥3g or 3 mL each) will be collected in clean containers at room temperature, fresh frozen at -20°C and then stored at -80°C within 72h. We will also obtain at colonoscopy four biopsies from inflamed and non-inflamed ileal and colonic mucosa (total 8 biopsies). From each individual, samples will be divided for analyses at Sheba and for transfer. Stool will be transferred to Prof. Elinav in Weizmann Institute to perform shotgun metagenomics of the microbiome. Intestinal biopsy and/or archived resection specimens (histology) will be transferred to Prof Stappenbeck at Washington University, St. Louis USA, for histological analysis of innate immune cells and paneth cell morphology analysis by H&E and immunohistochemistry.

Ileal and rectal biopsies will be collected and stored immediately in RNAlater. Biopsies will be obtained from each location (either inflamed or not inflamed, total 8 biopsies) and used for RNA and for microbial DNA extraction. RNA will be used for mRNAseq of tissue, and DNA for microbial characterization. mRNAseq will be done at the NIH supported digestive health center (DHC) core at Cincinnati Children Hospital Medical Center (CCHMC), where >700 mRNAseq of different IBD cohorts including RISK CD and PROTECT UC cohorts were already run with good results. Microbial 16S amplicon sequencing of stool & biopsy extracted DNA will be done as previously described.

Patients from both cohorts will also undergo environmental and dietary exposure survey. For environmental exposure, we will use the questionnaire developed by the International Organization of IBD (IOIBD), with some modification. The questionnaire consists of 87 questions covering 25 different topics proposed to be environmental risk factors for CD and/or UC. This questionnaire has been previously used in epidemiological studies investigating triggers of IBD, including one conducted in South-East Asia and China. Questions relate to five main different areas: (i) Childhood factors up to 20 years including breast feeding, appendectomy, tonsillectomy, eczema, vaccinations (tuberculosis, pertussis, measles, rubella, diphtheria, tetanus, polio), childhood infections (measles, pertussis, rubella, chickenpox, mumps, scarlet fever) and pet ownership; (ii) food habits including daily, weekly or less frequent consumption of fruit, vegetables, egg, cereal, bread, cereal, coffee, tea, juice, sugar and fast food; (iii) smoking habits (current smoker, non-smoker, ex-smoker); (iv) sanitary conditions such as the availability of in-house water tap, hot water tap or flush toilet; and (v) others factors including daily physical activity, oral contraceptive pill and stressful events before diagnosis. We will also add to the IOIBD questionnaire items pertaining to antibiotic use before and after the age of 15 years, use of toothpaste and presence of amalgam teeth filling during childhood or later in life.

For mapping dietary habits we will employ an interview conducted by a trained dietician and using the validated structured FFQ (Food frequency Questionnaire). This tool captures >600 food items, prioritized by their pre-defined frequency in regular diet. Personnel will be trained in the dietary interview method. FFQ results will be further imported into computerized FFQ version, which automatically derives and normalizes the nutrients content from an individual patient diet based on known Israel food-items nutrients' database from the National Institute of Statistics. As shown in the screen-shot figure from this responsive software for an exemplary patient, each color bar denotes a specific nutrient consumption by the individual (e.g protein, oligosaccharides, etc), along with its divergence from WHO normalized consumption (green colored range). The FFQ methodology will be complemented by a validation prospective three-day dietary itinerary capture by SmartPhone. Participants will take electronic pictures of all food items consumed during these three day. Photos will be uploaded to electronic visual data base, and food items will be identified, recorded and verified against the retrospective FFQ.

In order to prioritize among the multiple environmental/dietary factors, we will perform a systematic review and meta-analysis of all publications pertaining to environmental risk-factors for CD. We will compute pooled odds ratio and point estimates for each variable, and define the weighted effects between variables using random effect model. This will enable to dissect and identify factors which have been most reproducibly and robustly found to be associated with occurrence of CD. We will then prioritize these variables in a step-wise manner, for the analysis of environmental factors association with microbiome, transcriptome and PCP perturbations.

ELIGIBILITY:
Inclusion Criteria:

* adults>18YO
* CD patients: known CD\ new-onset CD\ travelling CD or controls: healthy individuals\ family members of CD patients

Exclusion Criteria:

* Age<18YO
* pregnant women
* inability to provide informed consent
* drug/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Correlation of microbiomic profile with dietary-environmental exposures in rural healthy population compared with urban healthy population in China and with new-onset Crohn's disease in Israel and China | A pilot study of 18 months
  Measurements: questionaries, physiological parameters (blood, stool, biopsies), inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel